CLINICAL TRIAL: NCT04143412
Title: Antiproteinuric Efficacy of ACE Inhibitors, Selective MRAs and ACE Inhibitor/Selective MRA Combination Therapy in Diabetic Hypertensives With Microalbuminuria
Brief Title: Efficacy of ACE Inhibitors, MRAs and ACE Inhibitor/ MRA Combination
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mostafa El Mokadem, Principal Investigator, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAAS blockers in albuminuria
Record Dates: First submitted 2019-10-26; First posted 2019-10-29 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Diabetic Nephropathy Type 2; Microalbuminuria Due to Type 2 Diabetes Mellitus
Keywords: microalbuminuria; Diabetic nephropathy; Hperkalemia; Eplerenone; Ramipril
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Ramipril; Eplerenone

STUDY DESIGN:
Intervention Model Description: Three parallel groups of therapy; Ramipril 10 mg monotherapy (25 patients) ,Eplerenone 50 mg monotherapy (25 patients) and combination therapy of Eplernone/Ramipril 50/10 mg (25 patients)
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tritace (Ramipril) (Active Comparator): 25 patients with type 2 diabetes mellitus and mild hypertension will be randomized to Tritace (Ramipril) 10 mg/ day. Full doses will be reached by forced titration after 4 weeks
  Interventions: Drug: Tritace (Ramipril 10 mg)
- Eraloner (Eplerenone) (Active Comparator): 25 patients with type 2 diabetes mellitus and mild hypertension will be randomized to Eraloner (Eplerenone) 50 mg/ day. Full doses will be reached by forced titration after 4 weeks
  Interventions: Drug: Tritace (Ramipril 10 mg)
- Tritace/Eraloner (Ramipril/Eplerenone)combination therapy (Active Comparator): 25 patients with type 2 diabetes mellitus and mild hypertension will be randomized to Tritace/Eraloner (Ramipril 10 mg / Eplerenone 50 mg ) / day. Full doses will be reached by forced titration after 4 weeks
  Interventions: Drug: Tritace (Ramipril 10 mg)

INTERVENTIONS:
Drug: Tritace (Ramipril 10 mg) — Stratified randomized clinical trial
  Other Names: Eraloner (Eplerenone 50 mg); Tritace/ Eraloner (Ramipril 10 mg/ Eplerenone 50 mg)

SUMMARY:
The aim of our work is to compare the antiproteinuric efficacy of ACEI monotherapy, Selective MRA monotherapy and their combination in mildly hypertensive patients with type 2 diabetes mellitus and microalbuminuria

DETAILED DESCRIPTION:
Diabetic nephropathy (DN) is the most common cause renal failure in Western countries, responsible for 45% of patients on renal replacement therapy.Diabetic nephropathy was characterized in the early stage by increased albumin excretion in urine, known as microalbuminuria. (DN) results from interactions between different pathological factors that include hyperglycemia, increased activity of the renin-angiotensin-aldosterone-system (RAAS), uncontrolled high systemic and glomerular pressure . (DN) optimal therapy continues to evolve. The main lines of treatment include strict glycemic and blood pressure (BP) control. The angiotensin converting enzyme (ACE) inhibitors have been known to reduce proteinuria both in normotensive and hypertensive patients with diabetic nephropathy and in hypertensive individuals with end stage renal failure . The mechanism by which ACE inhibitors exert their effect on proteinuria reduction is still unknown. The control of high systemic arterial pressure can be beneficial by reducing the filtration pressure. However, no association has been found between antihypertensive effect and proteinuria reduction in several studies. Microalbuminuria which is an early sign of nephropathy can be decreased also by use of Angiotensin receptor blockers (ARBs) in patients with type 2 diabetes mellitus . Insufficient blockade of aldosterone may lead to inadequate anti-albuminuric effects. Studies show that renin-angiotensin-aldosterone system inhibition with ACEI/ARB alone sometimes does not achieve optimal renoprotective effects and does not reduce progression of renal disease, despite therapy. Addition of mineralocorticoid receptor antagonists (MRAs) to angiotensin-converting enzyme inhibitor or angiotensin II receptor blocker therapy was found to reduce proteinuria in patients diabetic nephropathy and can delay progression of renal dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and non-pregnant female patients with established diagnosis of type 2 DM at least five years ago with glycosylated hemoglobin (HbA1c) ≤ 8.5%
* Age 30-80 Y
* Stage 1 hypertension (systolic BP 140-159 mmHg and/or diastolic BP 90-99 mmHg) and microalbuminuria diagnosed by measuring Urinary albumin/creatinine ratio (UACR) . Microalbuminuria was defined at a level between (30-300 mg/g)
* Patients included in our study had never been treated with ACEIs, ARBs or aldosterone antagonists, serum potassium level ≥ 3.5 and ≤ 5.0 mmol/L before randomization with estimated glomerular filtration rate (e GFR) ≥50 mL/min/1.73 m2

Exclusion Criteria:

* Patients with type 1 diabetes mellitus
* Patients with BP ≥ 160/100 mmHg
* Patients with secondary hypertension
* Non-diabetic nephropathy including (chronic glomerulonephritis, polycystic kidney disease and nephrosclerosis),
* Confirmed bilateral renal artery stenosis or stenosis of the renal artery in solitary functioning kidney
* History of New York Heart Association functional class III and IV heart failure
* Patients with rapid progression of kidney disease and women who were pregnant, breast-feeding, or planning to become pregnant during the study period

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Urinary albumin/creatinin ratio (UACR) | 24 weeks
  Percentage change in albumin/creatinin ratio compared with the baseline value

SECONDARY OUTCOMES:
Blood pressure | 24 weeks
  change in blood pressure level
estimated Glomerular Filtration Rate (e GFR) | 24 weeks
  change in estimated Glomerular Filtration Rate (e GFR)
Serum K | 24 weeks
  change in serum K level

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa O El Mokadem, M.D., Principal Investigator — Cardiology department,Faculty of Medicine, Beni-Suef University
Locations (1):
- Faculty of Medicine,Beni-Suef University, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No
To respect privacy and confidentiality of our patients

REFERENCES:
- [Background] Espinel E, Agraz I, Ibernon M, Ramos N, Fort J, Seron D. Renal Biopsy in Type 2 Diabetic Patients. J Clin Med. 2015 May 18;4(5):998-1009. doi: 10.3390/jcm4050998. PMID 26239461
- [Background] Zelmanovitz T, Gerchman F, Balthazar AP, Thomazelli FC, Matos JD, Canani LH. Diabetic nephropathy. Diabetol Metab Syndr. 2009 Sep 21;1(1):10. doi: 10.1186/1758-5996-1-10. PMID 19825147
- [Background] Cao Z, Cooper ME. Pathogenesis of diabetic nephropathy. J Diabetes Investig. 2011 Aug 2;2(4):243-7. doi: 10.1111/j.2040-1124.2011.00131.x. PMID 24843491
- [Background] Satirapoj B, Adler SG. Prevalence and Management of Diabetic Nephropathy in Western Countries. Kidney Dis (Basel). 2015 May;1(1):61-70. doi: 10.1159/000382028. Epub 2015 May 1. PMID 27536666
- [Background] Jalal S, Sofi FA, Abass SM, Alai MS, Bhat MA, Rather HA, Lone NA, Siddiqi MA. Effect of amlodipine and lisinopril on microalbuminuria in patients with essential hypertension: A prospective study. Indian J Nephrol. 2010 Jan;20(1):15-20. doi: 10.4103/0971-4065.62090. PMID 20535265
- [Background] Galle J. Reduction of proteinuria with angiotensin receptor blockers. Nat Clin Pract Cardiovasc Med. 2008 Jul;5 Suppl 1:S36-43. doi: 10.1038/ncpcardio0806. PMID 18580865
- [Background] Cagnoni F, Njwe CA, Zaninelli A, Ricci AR, Daffra D, D'Ospina A, Preti P, Destro M. Blocking the RAAS at different levels: an update on the use of the direct renin inhibitors alone and in combination. Vasc Health Risk Manag. 2010 Aug 9;6:549-59. doi: 10.2147/vhrm.s11816. PMID 20730071
- [Background] Cooper LB, Lippmann SJ, Greiner MA, Sharma A, Kelly JP, Fonarow GC, Yancy CW, Heidenreich PA, Hernandez AF. Use of Mineralocorticoid Receptor Antagonists in Patients With Heart Failure and Comorbid Diabetes Mellitus or Chronic Kidney Disease. J Am Heart Assoc. 2017 Dec 23;6(12):e006540. doi: 10.1161/JAHA.117.006540. PMID 29275368